CLINICAL TRIAL: NCT06643156
Title: A Multicenter, Open-label, Single-arm, Exploratory Clinical Study on the Tolerability, Safety and Efficacy of GP681 Powder for Oral Suspension in the Treatment of Uncomplicated Influenza in Pediatric and Adolescent Patients
Brief Title: Study to Assess the Tolerability, Safety and Efficacy of GP681 Powder for Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP681-S-202404
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GP681 powder for oral suspension 10mg/20mg/40mg (Experimental): All patients will receive a single oral dose of GP681 dry suspension dissolved in approximately 10 mL of warm water. The mixture will be stirred thoroughly before administration, and then the cup will be rinsed twice with an additional 10-20 mL of warm water (about 40°C) to ensure the full dose is taken.
  The dosage of GP681 in patients 2-18 years of age is a single weight-based dose displayed in the following table.
  Dosage Patients 40mg Aged 5-18years(exclusive)，weight≥40kg 20mg Aged 5-18years(exclusive)，20kg≤weight<40kg 40mg Aged 5-18years(exclusive)，20kg≤weight<40kg 10mg Aged 2-5years(exclusive)，10kg≤weight<20kg 20mg Aged 2-5years(exclusive)，10kg≤weight<20kg
  Interventions: Drug: GP681 10mg/20mg/40mg

INTERVENTIONS:
Drug: GP681 10mg/20mg/40mg — 0.5/1/2×20mg power for oral suspension taken orally

SUMMARY:
This study aims to evaluate the tolerability, safety, pharmacokinetic characteristics and efficacy of a single oral dose of GP681 powder for oral suspension in pediatric and adolescent patients with uncomplicated influenza. The study will also explore the optimal dose for a confirmatory clinical trial. Eligible patients who have been confirmed influenza virus infection and have experienced influenza symptoms within 48 hours prior to enrollment, will receive single dose of GP681 powder for oral suspension. The primary outcome measures included the observation of adverse events during the study, the pharmacokinetic parameters, as well as the efficacy endpoints including time to alleviation of influenza symptoms, viral clearance rate, changes in viral load, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 2 to 18 years (≥2 years and <18 years).
2. For participants aged 5 to 18 years (excluding 18 years): body weight ≥20 kg; for participants aged 2 to 5 years (excluding 5 years): 10 kg≤body weight <20 kg.
3. Diagnosed with influenza virus infection based on the following criteria: • Positive rapid antigen test (RAT) result from a throat or nasal swab for influenza virus (rapid nucleic acid tests or other rapid molecular diagnostic tests are also acceptable); and

   * Fever at screening (axillary temperature ≥37.5°C). If antipyretics have been administered, axillary temperature should be ≥37.5°C at least 1 hour after administration, or fever (axillary temperature <37.5°C) that returns to ≥37.5°C more than 4 hours after antipyretic use; and
   * At least one moderate or severe respiratory symptom at screening, including cough and/or nasal congestion or runny nose.
4. Time interval between the onset of illness symptoms and enrollment is ≤48 hours.

   Onset of illness: defined as the time of the first temperature increase (axillary temperature ≥37.5°C) or the time when at least one respiratory symptom related to influenza virus infection is first noticed by caregiver.
5. The participant's legal guardian agrees to the child's participation in the clinical study and signs the informed consent form (ICF). Participants aged ≥8 years must also voluntarily sign the ICF.
6. The investigator assesses that the participant and/or the caregiver can comply with the protocol requirements, follow-up visits, and complete all study procedures and evaluations, including diary card entries.

Exclusion Criteria:

1. Known allergy to the active ingredients or excipients of the investigational drug GP681.
2. Patients diagnosed with severe or critical influenza at screening: (1) Severe influenza cases were defined by the presence of one or more of the following conditions: a. Breathing difficulty and/or increased respiratory rate: >30 breaths/min for children >5 years old, >40 breaths/min for children aged 2-5 years; b. Consciousness alteration: slow response, somnolence, agitation, seizures, etc; c. Severe vomiting or diarrhea with moderate or severe dehydration; d. Pneumonia; e. Significant exacerbation of underlying diseases. (2) Critical influenza cases were defined by the presence of one or more of the following conditions: a. Respiratory failure; b. Acute necrotizing encephalopathy; c. Septic shock; d. Multiple organ dysfunction; e. Other severe clinical conditions requiring intensive care treatment.

   Note: Refer to the "Expert Consensus on Diagnosis and Treatment of Influenza in Children (2020 Edition)" for the criteria of severe/critical influenza.
3. History of any gastrointestinal disease known to affect drug absorption (including but not limited to gastroesophageal reflux disease, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, or post-gastrectomy conditions).
4. Suspected or confirmed bronchitis, pleural effusion, or interstitial pneumonia via clinical or radiological examination at screening.
5. Use of anti-influenza antiviral drugs within two weeks before screening (including neuraminidase inhibitors, hemagglutinin inhibitors, and M2 ion channel blockers such as oseltamivir phosphate, zanamivir, peramivir, favipiravir, arbidol, baloxavir, amantadine, or rimantadine, or other anti-influenza antiviral drugs approved by the NMPA).
6. Clinically relevant abnormal results in physical examination, 12-lead ECG, vital signs, hematology, clinical biochemistry, or urinalysis at screening, which in the investigator's judgment may pose a risk to the participant's safety, affect the study results, or impact the participant's ability to complete the study.
7. Acute respiratory tract infection, otitis media, or sinusitis within two weeks before screening.
8. Co-infection requiring systemic antibiotics or other systemic therapy at screening.
9. Known or suspected active primary or secondary immunodeficiency, including a history of HIV infection or other severe immunodeficiencies.
10. Known or suspected congenital abnormalities of the heart or lungs, or severe primary diseases affecting the cardiovascular, hepatic, renal, or hematopoietic systems, or evidence of active liver disease, including but not limited to jaundice or AST/ALT levels exceeding two times the upper limit of normal (ULN) at screening.
11. Positive serology for hepatitis B surface antigen or a history of hepatitis B infection at screening.

    Note: Children and adolescents with a history of hepatitis B vaccination without a history of hepatitis B infection do not need to be screened for this criterion (assessed via medical history).
12. Obesity as determined by the investigator: For participants <6 years old: BMI >97th percentile for the corresponding age and gender group; For participants ≥6 years old: BMI ≥obesity threshold for the corresponding age and gender group.

    Note: Refer to "WS/T 423-2022: Growth Standards for Children Under 7" or "WS/T586-2018: Screening for Overweight and Obesity in School-Aged Children and Adolescents."
13. History of mental illness, intellectual disability, substance abuse, or other adverse conditions (e.g., inability to read, understand, or write) that, in the investigator's judgment, may limit participation in the study.
14. Vaccination with an influenza vaccine within six months before screening or during the study period.

    Note: Participants' influenza vaccination history should be carefully reviewed before study enrollment (assessed via medical history).
15. Participation in a clinical trial of any investigational drug or device for any indication within 30 days prior to screening.
16. Intolerance to skin puncture, fainting at the sight of blood or needles, or poor venous access for blood collection at screening.
17. Other conditions judged by the investigator to be unsuitable for participation in the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to Day 15
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Time to Alleviation of Symptoms (TTAS) | up to Day 15
  Defined as the time from the treatment start to meeting both the following criteria (a and b), with all criteria maintained for at least 21.5 hours:
  a. Time from treatment initiation to the normalization of body temperature (axillary temperature ≤37.4°C).
Viral clearance rate on Day 2 and Day 5 (if applicable) | Days 2, 5
  Defined as the proportion of patients with viral titers below the quantifiable detection limit from the treatment start to Day 2 and Day 5 (if applicable)
Proportion of patients with influenza viral RNA positivity (by Q-PCR) and measurable viral titers at each time point (Day 2 and Day 5, if applicable) | Days 2, 5
  The percentage of patients positive for virus RNA by RT-PCR.Virus titer was quantified from nasopharyngeal swabs by tissue culture methods.
Area Under the Concentration (AUC) of virus RNA by RT-PCR and AUC of virus titer | Up to Day 5
  AUC of the viral load by RT-PCR and AUC of viral titer measured from baseline to Day 5
Change From Baseline in Virus RNA (RT-PCR) at Each Time Point | Days 2, 5
  Nasopharyngeal swabs were obtained for viral quantitation.
Time to Resolution of Fever | Up to Day15
  Defined as the time to a score of 0 (none) or 1 (mild) for individual symptoms from the 16 items on the CARIFS scale, sustained for at least 21.5 hours.
Time to return to normal activities of daily life | Up to Day15
  Defined as the time between the initiation of the study treatment and the return to normal activities of daily life.
Incidence of influenza-related complications | Up to Day15
  Defined as the percentage of subjects in the analysis population who experience each influenza-related complication (hospitalization, death, sinusitis, bronchitis, otitis media, and pneumonia) as an adverse event after the initiation of the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Women and Children's hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No